CLINICAL TRIAL: NCT04720495
Title: One-stage Versus Two-stage Inverted U-shaped Ridge Splitting With Simultaneous Implant Placement for Treatment of Anterior Maxillary Alveolar Ridge Undercut (a Comparative Randomized Clinical Trial)
Brief Title: One-stage Versus Two-stage Inverted U-shaped Ridge Splitting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hams Hamed Abdelrahman (Other)
Responsible Party: Sponsor-Investigator, Hams Hamed Abdelrahman, Assistant lecturer of DPH and Clinical statistician, Alexandria University
Organization: Alexandria University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Ridge_splitting
Record Dates: First submitted 2021-01-19; First posted 2021-01-22 (Actual); Last update posted 2021-01-22 (Actual); Status verified 2021-01

CONDITIONS: Maxillary Ridge Augmentation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- One stage ridge splitting (Active Comparator)
  Interventions: Procedure: One stage ridge splitting with simultaneous implant placement
- Two-stage ridge splitting (Experimental)
  Interventions: Procedure: Two-stage ridge splitting with implant placement

INTERVENTIONS:
Procedure: One stage ridge splitting with simultaneous implant placement — A full mucoperiosteal flap was raised using the sharp periosteal elevator to expose the bone crestally and buccally.
  An inverted U-shaped bone cut, down to the cancellous bone, was done in the undercut area with a piezoelectric device.
  The horizontal bone cut was made apical to the most concave point in the undercut area with a distance of 3 mm.
  The two vertical bone cuts were placed at least 1 mm away from the adjacent roots and extended beyond the undercut area.
  The released bone end was minimally elevated using a periosteotome through a greenstick fracture.
  All implants were installed with the implant shoulders flush to the bone level using a low-speed drilling procedure.
  Arms: One stage ridge splitting
Procedure: Two-stage ridge splitting with implant placement — The first surgery is the same as one stage ridge splitting Four weeks later, after revascularization between the bone block and the mucoperiosteum, the second surgery will be performed.
  A crestal incision was done and the envelope flap slightly elevated to preserve the blood supply.
  The implants will be placed in the same manner as one stage ridge splitting
  Arms: Two-stage ridge splitting

SUMMARY:
Fourteen patients having anterior maxillary undercut defect were selected to match a list of inclusion and exclusion criteria.

The participants were randomly allocated using a computer system into two groups:

Group A undergo inverted U-shaped maxillary ridge splitting using piezotomes with simultaneous implant placement in the same surgery.

Group B undergo inverted U-shaped maxillary ridge splitting as a first stage and after four weeks, ridge expansion and implant placement will be performed with only envelop flap.

Assessment included measurements of bone gain at the undercut defect and bone density labial to implants in each group from the cone-beam computed tomography

ELIGIBILITY:
Inclusion criteria

* Adult patients (20-45) years of age with no sex predilection
* At least one tooth missing in the anterior maxilla
* The presence of a labial undercut >2 mm in thickness which is not able to house an implant
* The presence of adequate bone width near the alveolar bone crest
* The absence of a vertical bone defect.

Exclusion criteria

* History of any systemic disease that would contraindicate surgery example uncontrolled diabetes.
* Pregnancy or lactation.
* Long-term amino-bisphosphonate therapy.
* Smoking more than 10 cigarettes per day.
* Alcohol or drug abuse.
* Uncontrolled periodontal disease.
* Active infection.
* Inadequate inter-incisal space.
* Bruxism or clenching.

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
Change in bone density buccal to the implant | baseline and 4 months
  Bone density was evaluated by CBCT
Change in bone width gain at the undercut area | baseline and 4 months
  Bone width gain was evaluated by CBCT

CONTACTS AND LOCATIONS:
Locations (1):
- Outpatient Clinic of Oral and Maxillofacial Surgery Department, Faculty of Dentistry, Alexandria University, Alexandria, Egypt